CLINICAL TRIAL: NCT04173091
Title: Risk Stratification in Patients With Severe Tricuspid Regurgitation: Insights From the TRicuspid Regurgitation rEgistry (TRuE)
Brief Title: Risk Stratification in Severe Treatment-naive, Tricuspid Regurgitation
Acronym: TRuE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alexander Lauten, Professor, Head of Cardiac catheterization Laboratory, Charite University, Berlin, Germany
Other Study IDs: TRuE012013
Record Dates: First submitted 2019-11-16; First posted 2019-11-21 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: tricuspid regurgitation, tricuspid valve, percutaneous treatment, right ventricle
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No Intervention — No Intervention planed

SUMMARY:
This registry is aimed to characterize patients with severe tricuspid regurgitation for the purpose of patient selection for interventional treatment and identify factors related to adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

Severe functional tricuspid regurgitation

Exclusion Criteria:

prior surgery or congenital heart diseases with involvement of the tricuspid valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe functional tricuspid regurgitation diagnosed echocardiographically.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year
  Mortality due to all causes
All-cause mortality | 5 years
  Mortality due to all causes
All-cause mortality | 10 years
  Mortality due to all causes

SECONDARY OUTCOMES:
Cardiovascular mortality | 1 year
  Mortality due to cardiovascular causes
Cardiovascular mortality | 5 years
  Mortality due to cardiovascular causes
Cardiovascular mortality | 10 years
  Mortality due to cardiovascular causes
Number of hospitalizations | 1 year
  Number of hospitalizations due to right heart failure
Number of hospitalizations | 2 years
  Number of hospitalizations due to right heart failure
Number of hospitalizations | 5 years
  Number of hospitalizations due to right heart failure
Number of hospitalizations | 10 years
  Number of hospitalizations due to right heart failure

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - Brunilda Alushi, Berlin
  - Contilia Heart and Vascular Centre, Essen
  - Department of Internal Medicine and Cardiology, Heart Centre Leipzig, Leipzig
  - German Heart Centre, Munich
- Rabin Medical Centre, Tel Aviv, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided